CLINICAL TRIAL: NCT02787707
Title: ٍEffect of Iranian Traditional Medicine Remedy Compared With Placebo on Chemotherapy Induced Nausea and Vomiting in Breast Cancer; a Double-blind Randomized Controlled Cross-over Clinical Trial
Brief Title: Effect of Iranian Traditional Medicine Remedy on Chemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sadegh Shokri, Ph.D candidate of Persian medicine, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MashhadUMS
Record Dates: First submitted 2016-05-19; First posted 2016-06-01 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Nausea; Vomiting
Keywords: Breast cancer; Traditional medicine; Chemotherapy Induced Nausea and Vomiting; Bunium Persicum; Rhus Coriaria
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms | interventions — Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Active Comparator): 2.7 grams Persumac powder (Iranian traditional medicine remedy composed from sumac and Bunium Persicum) every 8 hour from 24 hour before to fifth day after chemotherapy.
  Interventions: Drug: Persumac
- control (Placebo Comparator): 2.7 grams Lactose every 8 hour from 24 hour before to fifth day after chemotherapy.
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: Persumac — 2.7 grams Persumac powder (Iranian traditional medicine remedy composed from sumac and Bunium Persicum) every 8 hour
  Other Names: Sumac and black Zirah
  Arms: intervention
Drug: lactose — 2.7 grams Lactose every 8 hour
  Other Names: Lactose powder
  Arms: control

SUMMARY:
The main objective of this research is the role of the Persumac(an Iranian traditional remedy) on refractory Chemotherapy Induced Nausea and Vomiting (CINV) in breast cancer patients. Investigators assess effect of Persumac on the number/severity of nausea/ vomiting in acute and delayed phase.

DETAILED DESCRIPTION:
The study was a double-blind, placebo controlled, Cross-over clinical trial of Iranian traditional remedy (Persumac) on chemotherapy induced nausea and vomiting in breast cancer patients. From October 2015 to May 2016, sample selection continued to be until the full sample size.

Executive steps of study:

1. Among patients referred for breast cancer, to the oncology clinic in Imam Reza hospital in Mashhad University of Medical Sciences, an oncology referral center in the North East of Iran; patients included in study who had at least one chemotherapy session and remain at least three sessions of Their chemotherapy cycle and had inclusion criteria.
2. The initial assessment of patients (Run- in): Concurrent with the visit of patient for chemotherapy (the first session of her/his chemotherapy in this study); during interview, study questionnaire was delivered to patient. It took a full explanation of how to complete it and return the next session.
3. In the second session of chemotherapy (in study); after eligibility qualification and obtaining consent form, patients randomly allocated into intervention and control groups, In accordance with the study protocol, interventions take place. Questionnaire was delivered to the patient again.
4. (Wash out): Sixth day after the second session of chemotherapy until a day before the third session of chemotherapy determined as Wash out period.
5. In the third session of chemotherapy-in study, after obtaining the previous questionnaire, patient received cross over interventions. Questionnaire delivered to the patient again.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of breast cancer,
* Clinical diagnosis of chemotherapy induced nausea and vomiting resistant to conventional therapy.

Exclusion Criteria:

* Clinical diagnosis of hypersensitivity to Sumac or Bunium Persicum,
* Clinical diagnosis of digestion disorders,
* Clinical diagnosis of non chemotherapy induced nausea and vomiting,
* Milk allergy,
* Clinical diagnosis of bleeding diathesis,
* Clinical diagnosis of non-breast cancer.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of nausea and vomiting in acute phase | first 24 hour after chemotherapy
  number and severity of nausea and vomiting, acquired from questionnaire

SECONDARY OUTCOMES:
Frequency and Severity of nausea and vomiting in acute phase | Day 2-5 of chemotherapy
  number and severity of nausea and vomiting, acquired from questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nazari, Ph.D, Study Director — School of Persian and Complementary medicine, Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Department of Oncology, Imam Reza Hospital, Mashhad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Derived] Nazari M, Taghizadeh A, Bazzaz MM, Rakhshandeh H, Shokri S. Effect of Persian Medicine Remedy on Chemotherapy Induced Nausea and Vomiting in Breast Cancer: A Double Blind, Randomized, Crossover Clinical Trial. Electron Physician. 2017 Jan 25;9(1):3535-3543. doi: 10.19082/3535. eCollection 2017 Jan. PMID 28243404